CLINICAL TRIAL: NCT03339492
Title: Prospective, Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Safety and Efficacy of Pulsed Electromagnetic Field (PEMF) Therapy as an Adjunctive Treatment to Surgical Repair of Full Thickness Rotator Cuff Tears
Brief Title: PEMF as Adjunctive Treatment Following Surgical Repair of Full Thickness Rotator Cuff Tears
Acronym: RCStim
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim results suggested that the study was not adequately powered to achieve the primary endpoint: superiority in retear rate reduction in PEMF treatment versus placebo.
Sponsor: Orthofix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP-1604PSRC
Record Dates: First submitted 2017-10-31; First posted 2017-11-13 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Full-thickness Rotator Cuff Tear
Keywords: rotator cuff; PEMF; Pulsed Electromagnetic Field; Rotator Cuff Repair; adjunctive therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active PEMF (Active Comparator): Subjects have 2 out of 3 chance to get the active device which emits a pulsed electromagnetic field (PEMF) from the RCStim Model 1114 device (right and left side models available). Double-blind randomization.
  Interventions: Device: RCStim Model 1114
- Control/placebo PEMF (Sham Comparator): Subjects have a 1 out of 3 chance to get the control/placebo device which does not emit a pulsed electromagnetic field (PEMF) from the RCStim Model 1114 device (right and left side models available). Double-blind randomization.
  Interventions: Device: RCStim Model 1114

INTERVENTIONS:
Device: RCStim Model 1114 — Active device emits PEMF signal; placebo/control device does not emit PEMF signal
  Other Names: Orthofix rotator cuff soft tissue stimulator

SUMMARY:
The primary objective of this study is to prospectively determine, at 12 months post-surgical repair of full thickness rotator cuff tears, the safety and efficacy of treating full thickness rotator cuff repairs with pulsed electromagnetic fields (PEMF). The hypothesis states that exposure to a pulsed electromagnetic field (PEMF) following surgical repair of a full thickness rotator cuff tendon tear reduces tendon re-tear rates. The strength of the shoulder muscles and the levels of pain in subjects after surgical repair of their rotator cuff adjunctively treated with an active PEMF device will also be measured.

DETAILED DESCRIPTION:
This Clinical Investigation Plan (CIP) describes the prospective, randomized, double-blind, placebo controlled study to evaluate the safety and efficacy of Pulsed Electromagnetic Field (PEMF) therapy as an adjunctive treatment to surgical repair of full thickness rotator cuff tears.

Rotator cuff tears are common musculoskeletal injuries which often require surgical intervention. Unfortunately, post-repair prognosis is poor, and surgical repairs have been reported to fail in up to 94% of cases (Galatz et. al., 2004). Repaired tissue tends to be fibrotic, disorganized, and reattaches poorly to the bony insertion. To improve tendon-to-bone healing, many non-invasive therapeutic devices have been utilized post-operatively including therapeutic ultrasound and shock wave therapy (Lovric et. al., 2013; Springer and Badgett, 2015).

In orthopedics, the use of these non-invasive therapeutic devices has become increasingly popular during the post-operative recovery period in an effort to enhance tissue healing. These devices are relatively inexpensive and easily obtainable and relatively easy to use, and are especially enticing as they can be brought into the patient's home and do not require frequent visits to the clinic. Additionally, non-invasive therapeutic devices can be used for a variety of applications, including promoting tissue healing prior to surgical intervention or in lieu of surgical intervention all together. Although there are numerous advantages to using non-invasive therapeutic devices, their efficacy has not yet been maximized.

Based on the pre-clinical work presented (Tucker et. al., 2016; Huegel et. al., 2017), it is believed that pulsed electromagnetic fields may be an effective adjunctive treatment for patients who have undergone surgical repair of a torn rotator cuff.

ELIGIBILITY:
Inclusion Criteria:

1. Subject may be male or female between 21 years of age and 80 years of age at the time of consent.
2. Subject must have a repairable (≥1 and ≤ 5 cm in the AP direction) full thickness tear of either the supraspinatus tendon or both the supraspinatus and infraspinatus tendons, as determined by MRI and confirmed intra-operatively (pre-debridement) during the surgical repair of the rotator cuff using a calibrated probe.

   a. Subjects who do not meet this criterion will be considered screen failures.
3. This must be the first rotator cuff repair surgery on the study shoulder with the following exceptions:

   1. Previous repairs of the teres minor and/or the subscapularis muscles are permitted.
   2. Previous acromioplasties, decompressions, and clavicular fracture repairs are permitted.
   3. Concurrent acromioplasties, subacromial decompressions and/or distal clavicular excisions are permitted.
   4. Concurrent fracture repairs or reconstructions are NOT permitted.
   5. Biceps tenodesis or tenotomy (open or closed) are permitted.
4. Subject must not have used NSAIDs for one (1) week prior to surgery.
5. Subjects must agree NOT to use NSAIDS suring the first 6 weeks of the study. Low dose aspirin (81 mg) is permitted.
6. Subject must be willing and able to participate in post-operative physical therapy exercises.
7. Subject must be willing and able to follow all study procedures and return for all study visits.
8. Subject must have reliable access to any iOS device using iOS v.9.3 or later or an Android device with WiFi access for downloading the free device-specific app.
9. Subject must understand and be willing to sign the IRB-approved Informed Consent Document.

Exclusion Criteria:

1. Subject has a tear <1cm or >5cm in size measured intraoperatively, pre-debridement, using a calibrated probe.

   a. Subjects who do not meet this criterion will be considered screen failures.
2. Subject has a BMI > 45.
3. Subject has a pacemaker or defibrillator.
4. Subject is not able to or is unwilling to have an MRI on the study shoulder.
5. Subject requires assistive devices to walk such as crutches or walkers.
6. Subject has a rotator cuff tear in which the subscpularis tendon requires repair.

   a. Biceps tenodesis or tenotomy (open or closed) is allowed.
7. Subject has a Fuchs score grade of 3 for fatty infiltration on any of the rotator cuff muscles.

   Grade 1: Normal muscle, no or some fatty streaks Grade 2: Moderately pathologic muscle; more muscle than fat Grade 3: Advanced degeneration; as much muscle as fat or less muscle than fat
8. Subject has moderate to severe arthritis based on preoperative imaging or as judged at the time of arthroscopy.

   1. Pre-operative x-ray findings consistent with Grade 3 or Grade 4 glenohumeral arthritis, where the grades are defined as follows:

      Grade 1: doubtful narrowing of joint space and possible osteophytic lipping; Grade 2: definite osteophytes and definite narrowing of joint space; Grade 3: moderate multiple osteophytes and definite narrowing of joint space and some sclerosis and possible deformity of bone contour.

      Grade 4: bone on bone morphology
   2. Intra-operative exposed subchondral bone involving >= 50% of either the humeral head, glenoid or both.
9. Subject has a known collagen disorder such as, but not limited to, osteogenesis imperfecta (OI) or Ehlers-Danlos syndrome (EDS).
10. Subject has a known inflammatory or autoimmune connective tissue disease such as, but not limited to, gout affecting the shoulder, scleroderma, SLE, rheumatoid disease, or calcific tendonitis of the shoulder.
11. Subject has a metabolic bone disease such as Paget's disease or osteomalacia.

    a. Subjects with osteoporosis are not excluded from the study.
12. Subject has a deltoid defect, deltoid palsy or any other pseudoparalysis.
13. Subject has HIV, hepatitis, or has had an active malignancy in the past 5 years.
14. Subject has had previous rotator cuff repairs or repairs of the labrum.

    a. See Inclusion Criterion #3 for permitted surgeries.
15. Subject has a diagnosis of fibromyalgia or other chronic pain syndrome.
16. Subject has shoulder pain of unknown etiology.
17. Subject has an active or on-going neoplastic disease, except for benign skin cancer(s).
18. Subject has undergone administration, within the last 30 days, of any type of corticosteroid (with the exception of asthma medications and ophthalmic medications), antineoplastic, immunostimulation or immunosuppressive agent.
19. Subject is septic or has a local or systemic infection.
20. Subject has an admitted active substance abuse problem which includes recreational drugs and/or narcotics or a history of substance abuse where history is defined as "not under the care of a physician" for more than 5 years.

    a. Prescriptive medical marijuana is not permitted, including CBD oils.
21. Subject consumes more than 14 (men) or 7 (women) standard drinks (alcoholic units) per week where a drink equals a 12 oz. beer, or a 5 oz. glass of wine, or a 1.5 oz. shot of liquor.
22. Subject is currently seeking or receiving worker's compensation for this injury or for an injury that has occurred more than12 months prior to enrollment in this study or subjects who are currently in litigation or who have a history of litigation related to musculoskeletal diagnoses.
23. Subject has a major mental illnesses including major depression, bipolar disorder, schizophrenia or dementia that would prevent them from following the protocol and/or independently completeing the patient reported outcomes measures.
24. Subjects who have coexistent cervical spinal pathologies such as radiculopathies or myelopathies.
25. Subject has a mental or physical condition that would prevent tem from complying with the study protocol.
26. Subject has any other condition that, in the opinion of the investigator, would prevent them from completing the study.
27. Subject is a prisoner.
28. Subject has participated in another clinical trial within the last 90 days. a. The last study visit attended by the subject starts the 90 day window.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
retear rate | 12 months
  A reduction in retear rates in subjects adjunctively treated with PEMF compared with those treated with a placebo (inactive) RCStim PEMF device following surgical repair of full thickness rotator cuff tears.

SECONDARY OUTCOMES:
Muscle Strength | 12 months
  Strength to be measured using the IsoForceEvo2 dynamometer in subjects treated with PEMF treated and compared with subjects receiving the placebo/control PEMF device
Penn Shoulder Score | 12 months
  100 point scale with three subscales (pain, satisfaction, function) where a 12 pt increase in score with time after PEMF treatment is minimally clinically significant

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - The CORE Institute, Phoenix, Arizona
  - Stanford University, Redwood City, California
  - UCSF Orthopedics, San Francisco, California
  - Sabesan Orthopedics Research, Atlantis, Florida
  - Coastal Orthopedics and Sports Medicine, Bradenton, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Andrews Institute, Gulf Breeze, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Univ. of Maryland Dept of Orthopedics, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Univ of Michigan Orthopedic Sports Medicine Program, Ann Arbor, Michigan
  - Univ Orthopedics Associates at Great Neck, Great Neck, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Cincinnati Sports Medicine, Cincinnati, Ohio
  - Univ. of Pennsylvania Orthopedics, Philadelphia, Pennsylvania
  - The Rothman Institute, Philadelphia, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - South Carolina Sports Medicine and Orthopedics, North Charleston, South Carolina
  - The Campbell Clinic, Germantown, Tennessee
  - Deutsch Shoulder, Houston, Texas
  - Atlantic Orthopedics, Virginia Beach, Virginia
  - Jordan-Young Research Institute, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No